CLINICAL TRIAL: NCT00354250
Title: A Phase II Study of SB-715992 (NSC-727990, IND-70273) in Advanced Renal Cell Cancer
Brief Title: Ispinesib in Treating Patients With Metastatic or Unresectable Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02928; 14577A; N01CM62201 (NIH)
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Renal Cell Cancer; Stage III Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — ispinesib; CK0238273

ARMS (1):
- Treatment (ispinesib) (Experimental): Patients receive ispinesib (SB-715992) IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ispinesib

INTERVENTIONS:
Drug: ispinesib — Given IV
  Other Names: CK0238273; SB-715992

SUMMARY:
This phase II trial is studying how well ispinesib works in treating patients with metastatic or unresectable kidney cancer. Ispinesib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy of SB-715992 in patients with advanced renal cell cancer who have received at least one prior therapy. This will be achieved by a multi-center, single arm phase II study to evaluate the proportion of patients who achieve a complete or partial response with this agent.

SECONDARY OBJECTIVES:

I. To assess the overall survival. II. To assess the time to progression. III. To evaluate the qualitative and quantitative toxicities of this regimen.

OUTLINE: This is a multicenter study.

Patients receive ispinesib (SB-715992) IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed renal cell carcinoma which is metastatic (M1); histopathology is not restricted; patients with unresectable primary tumor (but MO) are also eligible
* Patients must have measurable disease; x-rays, scans or physical examinations used for tumor measurement must have been completed within 28 days prior to registration; x-rays, scans or physical examinations for non-measurable disease must have been completed within 42 days prior to registration
* Patients with metastatic disease who have a resectable primary tumor and are deemed a surgical candidate may have undergone resection and have recovered from surgery; at least 28 days must have elapsed since surgery and patient must have recovered from any adverse effects of surgery
* Patients must have discontinued therapy due to toxicity or demonstrated progression of disease following a minimum of one prior therapy; prior therapies may include: immunotherapy with either interferon (IFN) and/or Interleukin-2 (IL-2) or prior anti-angiogenesis agents; at least 28 days must have elapsed since the last treatment; patients must have recovered from any adverse effects of prior therapy
* Patients may have received prior radiation therapy; at least 21 days must have elapsed since completion of prior radiation therapy; patients must have recovered from all associated toxicities at the time of registration
* Patients may not have received prior tubule, DNA, or mitosis targeting agents for the treatment of renal cell carcinoma
* Patients must have a ECOG performance status of 0 - 2
* Pregnant or nursing women may not participate in this trial; women and men of reproductive potential must have agreed to use an effective contraceptive method; women of child-bearing potential must have a negative urine pregnancy test
* Patients with a history of brain metastases or who currently have treated or untreated brain metastases are not eligible; patients with clinical evidence of brain metastases must have a brain CT or MRI negative for metastatic disease within 56 days prior to registration
* Absolute granulocyte count (AGC) ≥ 1,500 cells/mm3, hemoglobin ≥ 9 mg/dl, and a platelet count ≥ 100,000 cells/mm3 within 14 days prior to registration
* Patients must have a total bilirubin < 2 mg/dl obtained within 14 days prior to registration
* Patients must have SGOT and SGPT =< 2.5 x institutional upper limit of normal within 14 days prior to registration
* Patients must have a serum creatinine =< 2.0 or a calculated creatinine clearance >= 40 mL/min for patients with creatinine levels above institutional normal; this must be obtained within 14 days prior to registration
* Patients must have a corrected QT interval less than 0.47 seconds
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* Prohibited medications; SB-715992 is a moderate to significant in vitro inhibitor of CYP3A4; the following lists of medications/substances are moderate to significant inhibitors/inducers of CYP3A4 that, if administered concomitantly with SB-715992, may alter study drug exposure; the use of these medications/ substances within 14 days (=< 6 months for amiodarone) prior to the administration of the first dose of SB-715992 through discontinuation from the study is prohibited

  * Inhibitors of CYP3A4:

    * Antibiotics: Clarithromycin, erythromycin, troleandomycin, rifabutin, rifapentine
    * Antifungals: itraconazole, ketoconazole, fluconazole (doses > 200 mg/day), voriconazole
    * Antidepressants: nefazodone, fluovoxamine
    * Calcium channel blockers: verapamil, diltiazem
    * Miscellaneous: amiodarone*, bitter orange
  * Use of amiodarone within 6 months prior to the administration of the first dose of SB-715992 is prohibited.
  * Inducers of CYP3A4:

    * Anticonvulsants: phenytoin, carbamazepine, phenobarbital, oxcarbazepine
    * Antibiotics: rifampin, rifabutin, rifapentine
    * Miscellaneous: St. John's Wort, modafinil
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to SB-715992
* Patients must not have any uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/ social situations that would limit compliance with study requirements
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy; therefore, HIV-positive patients receiving combination anti-retroviral therapy are not eligible because of possible pharmacokinetic interactions with SB-715992
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-05; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Response rate defined as the proportion of patients who achieve a complete or partial response with ispinesib evaluated per RECIST | Up to 4 years
  If the response rate is 30% or more, further study would be proposed based on the estimates produced in this trial. Will be presented along with 95% confidence intervals.

SECONDARY OUTCOMES:
Overall survival | Up to 4 years
  Will be presented in Kaplan-Meier plots and the median values of each (if reached) will be reported.
Time to progression | Up to 4 years
  Will be presented in Kaplan-Meier plots and the median values of each (if reached) will be reported.
Qualitative and quantitative toxicities of this regimen graded according to NCI CTCAE | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stadler, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States